CLINICAL TRIAL: NCT04093505
Title: Randomized Phase-III Study to Compare Two Schedules of Gemtuzumab Ozogamicin as Adjunct to Intensive Induction Therapy and to Compare Intensive Postremission Therapy Double Blinded With or Without Glasdegib in Older Patients With Newly Diagnosed AML
Brief Title: Gemtuzumab Ozogamicin in Induction and Glasdegib in Postremission Therapy in Patients With AML (Acute Myeloid Leukemia)
Acronym: GnG
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study turned out no longer feasible. End of Recruitment: 25.5.2022
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Prof. Dr. Richard F Schlenk, Head of NCT Trials Center and Clinical Trials Office Hematology/Oncology, University Hospital Heidelberg
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCT-2017-0537
Record Dates: First submitted 2018-10-30; First posted 2019-09-18 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — glasdegib

STUDY DESIGN:
Intervention Model Description: The two research questions are addressed in a 2 by 2 factorial design. Patients are upfront randomized for the two induction schedules (GO-147 versus GO-1, ratio 1:1) and for Glasdegib or Placebo (double blinded, ratio 1:1) as adjunct to consolidation therapy and as single agent 6 months maintenance therapy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GO147_G (Experimental): GO147: Induction therapy: Gemtuzumab Ozogamicin 3mg/m² on days 1,4 and 7
  _G: Consolidation & Maintenance therapy Glasdegib 100mg on days 4 to 27
  Interventions: Drug: Gemtuzumab Ozogamicin 147; Drug: Glasdegib
- GO147_P (Placebo Comparator): GO147: Induction therapy: Gemtuzumab Ozogamicin 3mg/m² on days 1,4 and 7
  _P: Consolidation & Maintenance therapy Placebo 100mg on days 4 to 27
  Interventions: Drug: Gemtuzumab Ozogamicin 147; Drug: Placebo Oral Tablet
- GO1_G (Experimental): GO1: Induction therapy: Gemtuzumab Ozogamicin 3mg/m² on day 1
  _G: Consolidation & Maintenance therapy Glasdegib 100mg on days 4 to 27
  Interventions: Drug: Gemtuzumab Ozogamicin 1; Drug: Glasdegib
- GO1_P (Placebo Comparator): GO1: Induction therapy: Gemtuzumab Ozogamicin 3mg/m² on day 1
  _P: Consolidation & Maintenance therapy Placebo 100mg on days 4 to 27
  Interventions: Drug: Gemtuzumab Ozogamicin 1; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Gemtuzumab Ozogamicin 147 — Induction therapy: Gemtuzumab Ozogamicin 3mg/m² on days 1,4 and 7
  Other Names: GO147
  Arms: GO147_G; GO147_P
Drug: Gemtuzumab Ozogamicin 1 — Induction therapy: Gemtuzumab Ozogamicin 3mg/m² on day 1
  Other Names: GO1
  Arms: GO1_G; GO1_P
Drug: Glasdegib — Consolidation & Maintenance therapy Glasdegib 100mg on days 4 to 27
  Other Names: _G
  Arms: GO147_G; GO1_G
Drug: Placebo Oral Tablet — Consolidation & Maintenance therapy Placebo 100mg on days 4 to 27
  Other Names: _P
  Arms: GO147_P; GO1_P

SUMMARY:
The study is a randomized phase III trial with a 2x2 factorial design with measurable residual disease and event-free survival as primary endpoints, respectively. Patients are upfront randomized for the two induction schedules (Gemtuzumab Ozogamicin (GO)-147 versus GO-1; ratio 1:1) and for Glasdegib or Placebo (double blinded, ratio 1:1) as adjunct to consolidation therapy and as single agent 6 months maintenance therapy. Chemotherapy backbone for induction therapy is standard 7+3 with cytarabine 200mg/m² continuously day 1 to day 7, daunorubicin 60mg/m² days 1, 2 and 3 and for consolidation therapy intermediate dose cytarabine (1g/m², bi-daily, days 1,2,3). The trial is designed to gain evidence of anti-leukemic activity of GO and Glasdegib in older patients with newly diagnosed acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed acute myeloid leukemia according to the 2016 WHO classification
* Genetic and immunophenotypic assessment in one of the central laboratories
* No prior chemotherapy for leukemia except hydroxyurea to control hyperleukocytosis (≤ 7 days)
* Age ≥ 60 years, no upper age limit
* ECOG performance status (ECOG PS) ≤ 2. See appendix 18.1
* Pregnancy and childbearing potential:

  * Non-pregnant and non-nursing women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within a sensitivity of at least 25 mIU/mL within 72 hours prior to registration ("Women of childbearing potential" is defined as a sexually active mature woman who has not undergone a hysterectomy or who has had menses at any time in the preceding 24 consecutive months).
  * Female patients of reproductive age must agree to avoid getting pregnant while on therapy.
  * WOCBP must either commit to continued abstinence from heterosexual intercourse or begin one acceptable method of birth control (IUD, tubal ligation, or partner's vasectomy) during study and 6 months after end of study/treatment. Hormonal contraception is an inadequate method of birth control.
  * Men must use a latex condom during any sexual contact with women of childbearing potential, even if they have undergone a successful vasectomy and must agree to avoid to father a child during study and 6 months after end of study/treatment
* Signed written informed consent
* Ability of patient to understand character and consequences of the clinical trial

Exclusion Criteria

* AML with PML-RARA or BCR-ABL1
* Patients with known active central nervous system leukemia (assessed clinically).
* Prior treatment with a smoothened inhibitor (SMOi) and/or hypomethylating agent for AML. (Treatment of a preceding MDS (myelodysplastic syndrome) with HMA is not an exclusion criterion.)
* Inadequate renal function: creatinine > 1.5 x upper normal serum level; estimated creatinine clearance ≤30 ml/min (calculated using the standard method for the institution).
* Inadequate liver function: ALT and AST ≥ 2.5 x ULN), total bilirubin ≥ 1.5 x ULN; Alkaline phosphatase ≥ 2.5 x ULN. Known liver cirrhosis or history of veno-occlusive disease (VOD) or history of Sinusoidal Obstruction Syndrome (SOS)
* Uncontrolled hypertension; severe obstructive or restrictive ventilation disorder
* Any one of the following ongoing or in the previous 6 months: myocardial infarction, congenital long QT syndrome, Torsades de pointes, arrhythmias (including sustained ventricular tachyarrhythmia), right or left bundle branch block and bifascicular block, unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure (CHF NYHA III/IV), cerebrovascular accident, transient ischemic attack or symptomatic pulmonary embolism; as well as bradycardia defined as <50 bpms
* QTc interval >470 msec using the Fredericia correction (QTcF).
* Uncontrolled infection
* Patients known to be refractory to platelet or packed red cell transfusions as per institutional guidelines, or who are known to refuse or who are likely to refuse blood product support.
* Patients with a "currently active" second malignancy other than non-melanoma skin cancer. Patients are not considered to have a "currently active" malignancy if they have completed therapy for more than one year and are considered by their physician to be at less than 30% risk of relapse within one year.
* Severe neurologic or psychiatric disorder interfering with ability of giving informed consent
* Known or suspected active alcohol or drug abuse
* Known positivity for HIV, active HBV, HCV, or hepatitis A infection
* Evidence or history of severe non-leukemia associated bleeding diathesis or coagulopathy
* No consent for biobanking and for registration, storage and processing of the individual disease-characteristics and course as well as information of the family physician about study participation.
* Pregnancy and lactation
* History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product
* Participation in a clinical study involving an investigational drug(s) (Phases 1-4) within 4 weeks prior to study entry.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
MRD-negativity | Collected during the first MRD-analysis after the first induction therapy cycle (after 4 weeks)
  Minimal Residual Disease negativity (MRD-negativity) after induction therapy measured by flow cytometry.

SECONDARY OUTCOMES:
EFS | Collected after 2 years follow-up time
  Event-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Heidelberg, Internal Medicine V, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jaramillo S, Krisam J, Le Cornet L, Kratzmann M, Baumann L, Sauer T, Crysandt M, Rank A, Behringer D, Teichmann L, Gorner M, Trappe RU, Rollig C, Krause S, Hanoun M, Hopfer O, Held G, Buske S, Fransecky L, Kayser S, Schliemann C, Schaefer-Eckart K, Al-Fareh Y, Schubert J, Geer T, Kaufmann M, Brecht A, Niemann D, Kieser M, Bornhauser M, Platzbecker U, Serve H, Baldus CD, Muller-Tidow C, Schlenk RF. Rationale and design of the 2 by 2 factorial design GnG-trial: a randomized phase-III study to compare two schedules of gemtuzumab ozogamicin as adjunct to intensive induction therapy and to compare double-blinded intensive postremission therapy with or without glasdegib in older patients with newly diagnosed AML. Trials. 2021 Nov 3;22(1):765. doi: 10.1186/s13063-021-05703-w. PMID 34732236